CLINICAL TRIAL: NCT06543472
Title: Dural Arteriovenous Fistulas Research at China INI
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XW0630
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dural arteriovenous fistula (DAVF) refers to abnormal connections between meningeal arteries and dural venous sinuses and/or subarachnoid veins. DAVF accounts for approximately 10% to 15% of intracranial vascular malformations. With advancements in imaging technology, increased awareness among physicians, and an aging population, the incidence of DAVF appears to be on the rise. Some literature even suggests it may surpass the occurrence of arteriovenous malformations. Several large-scale retrospective studies have been conducted internationally, involving over 1,000 cases, but some of their findings differ from what is commonly understood. Currently, there is a lack of large-sample single-center studies on DAVF, highlighting the urgent need for such research.

DETAILED DESCRIPTION:
Title：Dural Arteriovenous Fistulas Research at China INI.

Purpose：The incidence of DAVF is low. By collecting clinical data, we aim to establish a comprehensive database and biobank. This will help us elucidate the potential pathogenesis, vascular architecture, biological markers, and treatment outcomes of DAVFs. Furthermore, this study aims to address current controversies (such as treatment strategies for DAVF with pial arterial supply), unresolved issues (such as the optimal treatment and prognosis of infantile type DAVF), and further explore possible mechanisms of DAVF development.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with DAVFs who were admitted to Xuanwu Hospital.

Exclusion Criteria:

* Non-DAVF lesions confirmed by DSA.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All are from Chinese individuals.
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Long term prognosis | assessed at 3, 6, 12 and 24 months after procedure
  Safety endpoints include perioperative and postoperative complications, as well as the clinical status of the patients. This is evaluated using the preoperative modified Rankin Scale (mRS), mRS at discharge, and mRS at 6 to 12 months, along with the most recent clinical (inpatient/outpatient) or telephone follow-up. Efficacy endpoints include the immediate DAVF occlusion status after the last treatment, and the results from imaging follow-ups (DSA/MRA/CTA) at 6 to 12 months and the latest follow-up.

SECONDARY OUTCOMES:
Long-term cure rate | assessed at 3, 6, 12 and 24 months after procedure
  The recurrence rate of DAVF after confirmed complete cure, as determined by DSA/MRA/CTA

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Zhang, MD, Study Chair — Xuanwu Hospital Department of Neurosurgery; Xin Su, MD, Principal Investigator — Xuanwu Hospital Department of Neurosurgery; Zihao Song, MD, Principal Investigator — Xuanwu Hospital Department of Neurosurgery; Huiwei Liu, MD, Principal Investigator — Xuanwu Hospital Department of Neurosurgery; Peng Zhang, MD, Study Director — Xuanwu Hospital Department of Neurosurgery; Yongjie Ma, MD, Study Director — Xuanwu Hospital Department of Neurosurgery
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Su X, Li X, Song Z, Chen Y, Huang M, Liu H, Pang H, Zhang C, Sun L, Ye M, Hong T, Ma Y, Zhang H, Zhang P. Tentorial Dural Arteriovenous Fistulas: A Retrospective Cohort Study. Oper Neurosurg. 2025 Nov 1;29(5):678-685. doi: 10.1227/ons.0000000000001524. Epub 2025 Mar 5. PMID 40042314